CLINICAL TRIAL: NCT02296034
Title: Blood Glucose Variability in Obese Youth Participating in a Lifestyle Modification Program
Status: Withdrawn | Type: Observational
Why Stopped: Unable to recruit participants
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1409014604; K12DK094714 (NIH)
Record Dates: First submitted 2014-11-07; First posted 2014-11-20 (Estimated); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to measure blood glucose variation in youth prior to and after participation in a healthy lifestyle intervention program. The hypothesis is that youth with more severe obesity and those further along in puberty will have more glycemic variability, and that glycemic variability will be improved by participation in the lifestyle intervention program.

DETAILED DESCRIPTION:
Healthy lifestyle intervention programs aim to increase exercise and teach youth and about healthier dietary options, in hopes of avoiding obesity complications such as diabetes, and addressing the root causes of obesity. The program entitled Bright Bodies: A Lifestyle Intervention Program for Obese Youth, has been tested rigorously, showing significant improvements in body mass index and insulin resistance at both 1 and 2 years after the program and reversal of early abnormalities in glucose metabolism. While abnormalities on standardized oral glucose tolerance testing are well described in obese youth, this test may not reflect the "real life" glycemia changes in obese children. Understanding early glycemic changes in obese youth is important to better identify those at risk and strategize effective treatment plans, to avoid progression to prediabetes and diabetes. Thus the use of a continuous glucose monitor (CGM) may be a helpful adjunct to understanding the disease and therapy approaches in these patients.

A CGM is a device inserted under the skin on the abdomen which monitors glucose levels every 5 minutes, recording this information. CGM is commonly worn by kids with type 1 diabetes. The study will allow collection of information on glucose variability in much greater detail than can be seen from intermittent fingerstick glucose values or from an oral glucose tolerance test. Given the widespread epidemic of obesity and its complications, the ability to illustrate glycemic variability in obese youth is key to delineating risk categories and optimizing treatment. While lifestyle modification programs can be effective in improving measures of insulin sensitivity and OGTT results, their effect on real life glucose values has not been described. Hence the current study, aims to describe day-to-day glycemic variation in obese youth using CGM.

All enrolled subjects will wear a CGM for up to 7 days prior to initiation of the Bright Bodies program, and for up to 7 days at the end of the program. Additionally subjects will complete a food record and report exercise during both study periods. The study periods will take place during the 2 months prior to and the 2 months after completing the Bright Bodies program. The study will be explained to volunteers who meet eligibility criteria and informed consent/assent will be obtained. Demographic data will be recorded. Medical history will be obtained and a brief physical exam may be performed. Height, weight, BMI, percent body fat, fat mass, and fat free mass will be measured.

After enrollment subjects will meet with study personnel and learn how to keep a food record, with intermittent phone contact by study personnel to optimize food record compliance. They will also be asked to record exercise and any medications taken. A blinded CGM will be inserted at the beginning of each study period. Subjects will be educated regarding the CGM, including the requirement to measure blood glucose levels with a glucometer 3 times a day, at least every 12 hours (ideally on waking in the morning before eating, before dinner, and before bedtime), to calibrate the sensor. Subjects will be given a glucometer to obtain fingerstick blood sugar values and receive instruction regarding its use.

During the follow up visits the CGM will be removed, and the CGM and glucometer will be downloaded and collected. The food record will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Obese (BMI >95 percentile for age based on CDC growth charts)
* Willing to wear a CGM initially before and after the Bright Bodies program
* Willing to check fingersticks 3 times a day while wearing the CGM
* Willing to keep a food record before and after the Bright Bodies program
* Be in good general health without other acute or chronic illness that in the judgment of the investigator could interfere with the study or jeopardize subject safety
* Able to give consent (permission from parents and subject assent will be required)
* Female subjects of reproductive potential must be abstinent or consistently using appropriate family planning methods

Exclusion Criteria:

* Presence of any medical or psychiatric disorder that may interfere with subject safety or study conduct
* Prior participation in the Bright Bodies program.
* Diagnosis of diabetes
* Participation in a concurrent lifestyle modification (exercise/nutrition) program
* Use of any medications known to effect blood glucose levels, including oral or other systemic glucocorticoid therapy
* Subjects using herbal supplements will be excluded, due to the unknown effects of these supplements on glucose control
* Female subjects who are pregnant, lactating, or unwilling to be tested for pregnancy
* Subjects and/or parents who are not proficient in speaking/understanding the English language
* Subjects who discontinue participation in the Bright Bodies program during the study period will be excluded from follow-up monitoring

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Obese children participating in the Bright Bodies lifestyle intervention program
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2015-09 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in blood glucose pre and post meal | 4 months
  Change in blood glucose from meal time to 2-4 hours afterwards, before and after Bright Bodies program

SECONDARY OUTCOMES:
Change in mean number of calories consumed | 4 months
  Change in mean number of calories consumed before and after Bright Bodies program
Change in Glucose exposure | 4 months
  Change in glucose exposure as measured by the area under the curve before and after Bright Bodies program
Change in food consumption breakdown | 4 months
  Change in the percent of kcals from total fat, sugar, and protein of food consumed before and after Bright Bodies program

CONTACTS AND LOCATIONS:
Overall Officials: MIchelle Van Name, Principal Investigator — Yale University